CLINICAL TRIAL: NCT05293782
Title: The Effect of Trunk Kinesio Taping on Trunk Strength, Trunk Endurance, Balance and Plantar Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dilara Özen Oruk (Other)
Collaborators: Muğla Sıtkı Koçman University (Other)
Responsible Party: Sponsor-Investigator, Dilara Özen Oruk, Research Assistant, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 220001/23
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Trunk; Strength; Endurance; Plantar Pressure
Keywords: Taping; Body structure; muscle facilitation; postural stability

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Kinesiotaping on trunk flexor muscles (Active Comparator): Kinesiotaping
  Interventions: Other: Kinesitaping
- Kinesiotaping on trunk extensor muscles (Active Comparator): Kinesiotaping
  Interventions: Other: Kinesitaping
- Placebo Kinesiotaping on trunk flexor muscles (Placebo Comparator): Kinesiotaping
  Interventions: Other: Kinesitaping
- Placebo Kinesiotaping on trunk extensor muscles (Placebo Comparator): Kinesiotaping
  Interventions: Other: Kinesitaping

INTERVENTIONS:
Other: Kinesitaping — Kinesiotaping - muscle facilitation technique

SUMMARY:
This study perform to investigate the the acute effects of trunk kinesiotaping on trunk strength, trunk endurance, balance and plantar pressure.

DETAILED DESCRIPTION:
Body; It is an integral part of the body for spinal stability, postural control, proprioceptive stimuli, and energy transfer between the upper and lower extremities. Increasing trunk muscle endurance, strength and proprioception; It is of great importance in body function.

In this study, kinesiotape will apply to the trunk flexsor and extensor muscles using the muscle facilitation techniques. Also placebo taping will apply on the same muscles with same kinesiotape without any stretching or positioning. A total of 4 applications including kinesiotaping and placebo taping will perform randomly in 4 consecutive days.

For each subject; A total of 5 separate evaluations will perform on the first day (without taping) and following 4 consecutive days. Between the taping and evaluation of the subjects will wait for 30-45 minutes.

The aim of the study is to determine the effect of kinesio taping (KB) applied to different trunk muscles on various parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form and participated in all stages of the study
2. Being in the age range of 18-30

Exclusion Criteria:

1. Having any physical, mental or psychological illness that may affect participation in the study
2. Having an allergy to kinesio tape
3. Having a history of major surgery in the last six months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
A kinesthetic ability trainer (Sport KAT Model 650-TS) which shows the balance index scores | Change of balance from baseline at the end of 30 minutes of each kinesiotaping intervention.
  Change of static and dynamic balance
Diagnostic Support Electronic Baropodometry and Milletrix software | Change of plantar pressure from baseline at the end of 30 minutes of each kinesiotaping intervention.
  Change of plantar pressure
Back Leg Chest Dynamometer | Change of trunk muscles strength from baseline at the end of 30 minutes of each kinesiotaping intervention.
  Change of trunk muscles strength
Trunk muscles endurance tests (Modifiye Biering-Sorensen test, trunk flexion endurance test, lateral bridge test, plank test) | Change of trunk muscles endurance from baseline at the end of 30 minutes of each kinesiotaping intervention.
  Change of trunk muscles endurance

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Sıtkı Koçman University, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided